CLINICAL TRIAL: NCT03396744
Title: Bright Light Therapy in the Treatment of Non-seasonal Bipolar Depressive Episode of Bipolar Disorder: A Dose Research Phase I/II Trial
Brief Title: Bright Light Therapy in the Treatment of Non-seasonal Bipolar Depression
Acronym: LUBI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC16142
Record Dates: First submitted 2018-01-02; First posted 2018-01-11 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Dose finding study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning group (Active Comparator): Exposition at 8 a.m +/- 30 min, during 10 active weeks, and assessed 6 months after this intervention
  Interventions: Device: Light
- Mid-day group (Active Comparator): Exposition at 8 a.m +/- 30 min, during 10 active weeks, and assessed 6 months after this intervention.
  Interventions: Device: Light

INTERVENTIONS:
Device: Light — Placebo light (50 Lux) during 1 week and then active bright light with glasses using a dosage escalation (inter- and intra-subject) of 7.5, 10, 15, 30 and 45 min

SUMMARY:
Bipolar disorder (BD) is a severe brain disorder characterized by the recurrence of mood episodes. Depressive episodes in BD are frequently refractory and clinicians have few treatment options. Bright light therapy (BLT, also named phototherapy) is a promising emerging antidepressant strategy that is lacking evidence-based guidelines for its prescription in BD, including to avoid side effects such as manic switches. In this context, this study aimed to evaluate modalities of the BLT dosage (time of exposure) escalation depending on the tolerance (manic symptoms) in two groups exposed either during the morning or at mid-day.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a severe brain disorder characterized by the recurrence of mood episodes. Patients presenting with BD spend more time with depressive symptoms than with manic ones, which have a major impact on the quality of life and is associated with poorer outcomes including recurrences and suicide. In addition depressive phases in BD are frequently refractory and clinicians have few treatment options. Bright light therapy (BLT, also named phototherapy) is the first line treatment for depression with seasonal patterns and show promising results in the treatment of non-seasonal depressions. More evidence in non-seasonal depressions is expected, especially in BD. Moreover, some specificities linked to BD, such as the manic switch, warrant evidence-based therapeutic guidelines and so deserve more studies in BD. Preliminary reports suggest that morning exposure may induce manic switches, and that mid-day exposures may be associated with a decreased risk of manic switch. Different dose-titration protocols have also not been compared, and data are lacking. In this context, this study aimed to evaluate modalities of the BLT dosage (time of exposure) escalation depending on the tolerance (manic symptoms) in two groups exposed either during the morning or at mid-day.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged from 18 to 55 year-old.
* Patients must read and understand French language, and must provide written informed consent.
* Patients must be inpatients or outpatients followed in psychiatry for a major depressive episodes.
* Patients must have a diagnosis of bipolar disorder, type I or II, according to the DSM-5 and determined by a SCID.
* Patients must have a major depressive episode, at least of moderate intensity, according to the DSM-5, with a MADRS total score ≥20 and determined by a SCID.
* Patients must have a mood stabilizer since at least 4 weeks at standard dosage (lithium, or sodium valproate, or second generation antipsychotics such as quetiapine, aripiprazole, olanzapine).
* Female patients must be using a medically accepted means of contraception.
* Patients must be affiliated to the social security scheme.

Exclusion Criteria:

* Patients under guardianship or deprivation of liberty by administrative or judicial decision
* Seasonal pattern of major depressive episode according to DSM-5 criteria.
* Psychotic, mixed, or catatonic characteristics according to DSM-5 criteria
* High suicidal risk assessed by the Columbia Scale of Suicide Risk Severity (C-SSRS)
* Not stabilized comorbidities (addictive disorders according to the DSM-5 criteria or other decompensated general medical cause).
* Ophthalmic pathology (cataract, macular degeneration, glaucoma, retinitis pigmentosa) and diseases affecting the retina (retinopathy, diabetes, herpes, etc.).
* Photosensitive treatment, including the following treatments:

  * Cyclins (Vibramycin®, Doxycycline®)
  * Amiodarone (Cordarone®, Amiodarone®)
  * Phenothiazines (Largactil®, Modecate®, Nozinan®, Melleril®, Trilafon®)
  * Methotrexate (Methotrexate®)
  * Sulfamides (antibiotics, diuretics or hypoglycemic agents)
  * Chloroquine (Nivaquine®)
  * Some anti-inflammatories (Apranax®, Indocid®)
  * Psoralens used in puvatherapy
  * Isotretinoin (Roaccutane® and generics)
  * Verteporfin (Visudyne®).
* Lactating or pregnant women (pregnancy urine positive test).
* Subjects who have already used light therapy in the last 6 months.
* Therapeutic resistance of the current major depressive episode (≥2 traditional antidepressants such as SSRI, IRSNA, MAOI or tricyclic, at effective therapeutic dosage for more than 6 weeks)
* Use of another antidepressant strategy than the mood stabilizer, including antidepressants of all classes (which will have to be stopped before the initiation of light therapy) and psychotherapy with onset <1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in Mania Score | 10 weeks
  The Young Mania Rating Scale (YMRS) will be used as a measure of tolerance reflecting change in YMRS total scores at each week over the 10 weeks (Total score ≥ 12 defining an hypomanic switch).

SECONDARY OUTCOMES:
Change in Depression Score | 6, 8 and 10 weeks
  The Montgomery-Asberg Depression Rating Scale (MADRS) will be used as a measure of efficacy reflecting changes from baseline to endpoint
Change in Clinical Global Impressions (CGI) | 6, 8 and 10 weeks
  The Clinical Global Impressions (CGI) will be used as a measure of efficacy reflecting changes from baseline to endpoint
Change in tolerance | 1, 2, 3, 4, 5, 6, 8 and 10 weeks
  YMRS will be used to evaluate hypomanic switch at 3 days after each duration of exposition change
Acceptability | 1, 2, 3, 4, 5, 6, 8 and 10 weeks
  measured by auto-questionnaire made by the investigators
MADRS | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then at 6 months
  The MADRS will be used to evaluate changes of depressive symptoms from baseline
Clinical Global Impressions (CGI). | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then 6 months
Columbia-Suicide Severity Rating Scale (C-SSRS) | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then 6 months
Quick Inventory of Depressive Symptomatology (QIDS SR-16) | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then 6 months
Altman Self-Rating Mania Scale (ASRM). | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then 6 months
Pittsburgh Sleep Quality Index (PSQI). | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then 6 months
Composite Scale of Morningness (CSM). | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then 6 months
Circadian Type Inventory (CTI). | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then 6 months
Epworth Sleepiness Scale (ESS). | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then 6 months
Side effects: PRISE-M | 1, 2, 3, 4, 5, 6, 8 and 10 weeks, and then 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fenand Widal hospital, Paris, France

REFERENCES:
- [Derived] Geoffroy PA, Chevret S, Mauries S, Chaffaut C, Amad A, Bellivier F, Benard V, Courtet P, Dubertret C, Gorwood P, Mazer N, Mekaoui L, Olie E, Pataud G, Vaiva G, Lejoyeux M, Sit D, Maruani J. Bright Light Therapy in the Morning or Midday for the Treatment of Nonseasonal Depression in Bipolar Disorder (LuBi): A Dose-Escalation Phase 1/2 Randomized Double-Blind Trial. J Clin Psychiatry. 2025 Jun 23;86(3):25m15826. doi: 10.4088/JCP.25m15826. PMID 40608475
- [Derived] Geoffroy PA, Abbassi EMBE, Maruani J, Etain B, Lejoyeux M, Amad A, Courtet P, Dubertret C, Gorwood P, Vaiva G, Bellivier F, Chevret S. Bright Light Therapy in the Morning or at Mid-Day in the Treatment of Non-Seasonal Bipolar Depressive Episodes (LuBi): Study Protocol for a Dose Research Phase I / II Trial. Psychiatry Investig. 2018 Dec;15(12):1188-1202. doi: 10.30773/pi.2018.09.27.1. Epub 2018 Nov 26. PMID 30466205